CLINICAL TRIAL: NCT07355738
Title: A Randomized, Open-label, Single-dose, Parallel Comparison Study to Evaluate the Bioequivalence of GZR18 Injection Before and After CMC Change in Healthy Adult Male Subjects
Brief Title: Bioequivalence Study of GZR18 Injection Before and After CMC Change
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GZR18-OOO-108
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obesity&T2D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GZR18 injection A1 (Experimental): Single dose, s.c.
  Interventions: Drug: GZR18 injection A
- GZR18 injection B1 (Experimental): Single dose, s.c.
  Interventions: Drug: GZR18 injection B
- GZR18 injection A2 (Experimental)
  Interventions: Drug: GZR18 injection A
- GZR18 injection B2 (Experimental)
  Interventions: Drug: GZR18 injection B
- GZR18 injection A3 (Experimental)
  Interventions: Drug: GZR18 injection A
- GZR18 injection B3 (Experimental)
  Interventions: Drug: GZR18 injection B

INTERVENTIONS:
Drug: GZR18 injection A — Administered SC
  Arms: GZR18 injection A1; GZR18 injection A2; GZR18 injection A3
Drug: GZR18 injection B — Single dose, s.c.
  Arms: GZR18 injection B1; GZR18 injection B2; GZR18 injection B3

SUMMARY:
This is an open-label, randomized, single-dose, parallel comparison bioequivalence study conducted in healthy adult male subjects.

The study is divided into 3 parts, each of which evaluates the bioequivalence of GZR18 Injection for one strength before and after CMC changes.

Subjects eligible for each part of the screening will be randomized into Group A or Group B in a 1:1 ratio. Each subject will receive a single dose of GZR18 Injection, followed by PK blood sampling and safety follow-up for 35 days. Subjects will be admitted to the hospital 1 day predose, follow a standardized light diet that evening, and then fast for at least 10 h thereafter. On the day of administration, GZR18 Injection of a single strength will be administered subcutaneously under fasting conditions at a site approximately two finger-widths (2.5 cm) away from the umbilicus on the abdomen. Lunch and dinner will be served approximately 3 and 9 h postdose, respectively.

Venous blood will be collected at 14 time points for GZR18 plasma concentration analysis: at 0 h (within 60 min predose) and 1, 6, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, and 840 h postdose.

Subjects will undergo corresponding laboratory safety tests at screening, D36, and early withdrawal visits.

During the entire study period, subjects should maintain a light diet, avoid strenuous exercise, and refrain from consuming juice, caffeinated beverages (such as tea and coffee), and alcoholic drinks. Smoking and any other activities that may affect PK observation or safety evaluations are strictly prohibited.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily sign the Informed Consent Form (ICF), can receive SC injection, fully understand the content, process and possible adverse reactions of the trial, and are able to follow the regulations on contraindications and restrictions specified in this protocol.
2. Male, 18 to 50 years of age at signing the ICF (both inclusive).
3. Weight ≥ 50 kg and body mass index (BMI) within 19-26 kg/m2 (inclusive) at screening.
4. Subjects of childbearing potential with no birth plan from the signing of ICF to 8 weeks after the last dose, willingness to take effective contraceptive measures, and no plan for sperm donation.

   -

Exclusion Criteria:

1. Subjects with clinically significant abnormalities detected during the screening period in physical examination, vital signs, laboratory tests, 12-lead ECG, abdominal ultrasound, or chest X-ray, as determined by the investigator.
2. Subjects who test positive for hepatitis B virus surface antigen, hepatitis C virus IgG antibody, human immunodeficiency virus antibody, P24 antigen, or anti-treponema pallidum antibody.
3. Subjects with a history of or existing circulatory, urinary, digestive, respiratory, nervous, endocrine, or psychiatric disorders that, in the investigator's judgment, remain clinically significant.
4. History of acute or chronic pancreatitis and pancreatic injury before screening.
5. History or family history of previous or existing medullary thyroid carcinoma, multiple endocrine neoplasia type 2.
6. Subjects who have used any drugs that alter the activity of drug metabolizing enzymes or transporters within 4 weeks prior to screening, or subjects with acute diseases or concomitant medication from the screening period to before randomization.
7. Subjects with severe infection or unexplained infection within 4 weeks before screening.
8. Major surgery within 6 months prior to screening, or scheduled surgery or hospitalization during the study.
9. Subjects known or suspected to have hypersensitivity to any ingredient of the investigational medicinal product (IMP) (glucagon like peptide-1 receptor agonist (GLP-1RA) or its excipients).
10. Use of any prescription drugs, over-the-counter drugs or Chinese herbal medicine within 2 weeks prior to screening; use of any GLP-1R agonists or drugs with the same mechanism of action to GLP-1R agonists (such as GLP-1R/glucagon receptor [GCGR] agonists or gastric inhibitory polypeptide receptor [GIPR]/GLP-1R agonists or GIPR/GLP-1R/GCGR agonists) within 3 months prior to screening.
11. Subjects who have been vaccinated within 1 month before screening or are scheduled for vaccination during the study.
12. Blood donation or blood loss greater than or equal to 400 mL within 3 months before screening, or blood donation scheduled during the study or within 8 weeks after the end of the study.
13. History of drug abuse prior to screening; or positive results for drug abuse at screening (D-1).
14. History of alcohol abuse within 3 months prior to screening, defined as an average intake of more than 14 units per week (1 standard unit=360 mL of beer or 150 mL of 12% wine or 45 mL of 40% spirits); or use of any alcohol-containing products 48 hours before administration; or abnormal results for breath alcohol test at screening (D-1).
15. Subjects who smoked more than 5 cigarettes per day on average within the 3 months before screening, or who do not agree to abstain from smoking for the duration of the study.
16. Subjects who engage in strenuous exercise within 48 h before administration of the IMP, or have other factors that may affect drug absorption, distribution, metabolism, or excretion.
17. Subjects who consume grapefruit or grapefruit-containing products, or any caffeinated or xanthine-containing foods or beverages (such as coffee, tea, cola, or chocolate) within 48 hours before administration of the IMP.
18. Subjects who have special dietary requirements and cannot adhere to a standardized diet, or who are lactose intolerant.
19. Subjects with a history of needle phobia and blood phobia, difficulty in blood collection or intolerance to venous blood collection.
20. Subjects who are investigators or employees of the study site, or family members of the employees or investigators.
21. Participation in a clinical study of another IMP or device within 3 months before screening, or within 5 half-lives of the previous IMP (whichever is longer). Or plan to participate in another clinical study of an IMP or device before completing all scheduled assessments in the clinical study.

    -

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
the maximum concentration (Cmax) | Day1-Day36
the area under the concentration-time curve during a dosing interval (AUC0-t) | Day1-Day36
the area under the concentration-time curve from the time of dosing extrapolated to infinity (AUC0-∞) | Day1-Day36

SECONDARY OUTCOMES:
AUC extrapolated from the last time point extrapolated to infinity in percentage of the AUC0-∞ (AUC_%Extra) | Day1-Day36
time of maximum observed concentration (Tmax) | Day1-Day36
elimination half-life (t1/2) | Day1-Day36
elimination rate constant of plasma concentration at terminal phase (λz) | Day1-Day36
Treatment-Emergent Adverse Events (TEAEs) | Day1-Day36

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Suzhou, China